CLINICAL TRIAL: NCT00953680
Title: An Open-Label, Randomized, 2-Period Crossover Study to Evaluate the Bioequivalence After Administration of a Losartan 100-mg/Hydrochlorothiazide 12.5-mg Combination Tablet and the Coadministration of a Currently Marketed COZAAR™ 100-mg Tablet and MICROZIDE™ 12.5 mg Capsule in Healthy Adults
Brief Title: Bioequivalence of Losartan and Hydrochlorothiazide (HCTZ) Combination Tablet and Coadministration of Its Components (0954A-306)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-306; 2009_628
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2010-07-16 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination; Losartan; Hydrochlorothiazide

ARMS (2):
- losartan /HCTZ combination tablet (Active Comparator): single dose losartan 100 mg/HCTZ 12.5 mg combination tablet
  Interventions: Drug: losartan potassium (+) hydrochlorothiazide (HCTZ)
- losartan tablet + HCTZ capsule (Active Comparator): Single dose losartan 100 mg tablet + HCTZ 12.5 mg capsule
  Interventions: Drug: losartan potassium; Drug: hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Drug: losartan potassium (+) hydrochlorothiazide (HCTZ) — Single dose losartan 100 mg/HCTZ 12.5 mg combination tablet in one of two treatment periods.
  Arms: losartan /HCTZ combination tablet
Drug: losartan potassium — Single dose losartan 100 mg tablet in one of two treatment periods.
  Other Names: COZAAR™
  Arms: losartan tablet + HCTZ capsule
Drug: hydrochlorothiazide (HCTZ) — Single dose HCTZ 12.5 mg capsule in one of two treatment periods.
  Other Names: MICROZIDE™
  Arms: losartan tablet + HCTZ capsule

SUMMARY:
This study will evaluate the bioequivalence of the losartan/hydrochlorothiazide (HCTZ) combination tablet and coadministration of losartan and hydrochlorothiazide.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female between the ages of 18 and 45 years of age
* Subject does not smoke

Exclusion Criteria:

* Subject has a history of any illness that might pose additional risk to participation or confound the results of the study
* Subject has a history of hepatitis B or C or significant drug allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2004-04; Primary Completion 2004-05 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan-HCTZ Combination Tablet/Losartan Tablet +HCTZ Capsule: Single dose losartan 100 mg and hydrochlorothiazide (HCTZ) 12.5 mg combination tablet then a single dose losartan 100 mg tablet + HCTZ 12.5 mg capsule
- Losartan Tablet +HCTZ Capsule/Losartan-HCTZ Combination Tablet: Single dose losartan 100 mg tablet + hydrochlorothiazide (HCTZ) 12.5 mg capsule then a single dose losartan 100 mg and HCTZ 12.5 mg combination tablet
Period: Period 1
Arm/Group | Losartan-HCTZ Combination Tablet/Losartan Tablet +HCTZ Capsule | Losartan Tablet +HCTZ Capsule/Losartan-HCTZ Combination Tablet
Started | 38 | 39
Completed | 38 | 38
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Losartan-HCTZ Combination Tablet/Losartan Tablet +HCTZ Capsule | Losartan Tablet +HCTZ Capsule/Losartan-HCTZ Combination Tablet
Started | 38 | 38
Completed | 38 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized patients
Arm/Group | All Participants
Number analyzed (Participants) | 77
Age, Continuous [Mean (Full Range); unit: years] | 33.87 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 31
Height [Mean (Full Range); unit: Centimeters] | 166.81 [152 to 191]
Weight [Mean (Full Range); unit: kilograms] | 73.01 [50 to 99.1]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC(0 to Infinity)) of Losartan
Time Frame: 0 to 36 Hours Post Dose
Population: Pharmacokinetic (PK) results included complete data from 75 of 77 subjects (with 1 replacement). Partial data from 1 subject were not analyzed. Plasma concentrations for another subject were undetectable following 1 treatment, with partial data excluded from analyses.
Measure: Least Squares Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Losartan-HCTZ Combination Tablet: single dose losartan 100 mg and HCTZ 12.5 mg combination tablet
Arm/Group | Losartan-HCTZ Combination Tablet | Losartan Tablet + HCTZ Capsule
Number analyzed (Participants) | 75 | 75
ng*hr/mL | 1018.1 (382.5) | 1024.9 (354.6)
Statistical Analysis 1: Comparison: Losartan-HCTZ Combination Tablet vs Losartan Tablet + HCTZ Capsule; Least-Squares Mean Ratio (A/B); A= Single dose losartan 100 mg-HCTZ 12.5 mg combination tablet; B= Single dose losartan 100 mg tablet + HCTZ 12.5 mg capsule; Test type: Non-Inferiority or Equivalence — Equivalence Bounds of (0.80, 1.25); Least-Squares Mean Ratio = 0.993, 90% CI [0.950 to 1.039]

2. Primary Outcome: Peak Plasma Concentration (Cmax) for Losartan
Description: Peak Plasma Concentration (Cmax), or maximal concentration of drug following dosing.
Time Frame: 36 Hours Post Dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Losartan-HCTZ Combination Tablet | Losartan Tablet + HCTZ Capsule
Number analyzed (Participants) | 75 | 75
ng/mL | 532.7 (334.9) | 637.9 (425.3)
Statistical Analysis 1: Comparison: Losartan-HCTZ Combination Tablet vs Losartan Tablet + HCTZ Capsule; Least-Squares Mean Ratio (A/B); A= Single dose losartan 100 mg-HCTZ 12.5 mg combination tablet; B= Single dose losartan 100-mg tablet + HCTZ 12.5 mg capsule; Test type: Non-Inferiority or Equivalence — Equivalence Bounds of (0.80, 1.25); Least-Squares Mean Ratio = 0.835, 90% CI [0.749 to 0.931]

3. Primary Outcome: Area Under the Curve (AUC(0 to Infinity)) of HCTZ
Description: Plasma Area Under the Curve, a measure of drug exposure following dosing
Time Frame: 0 to 30 Hours Post Dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Losartan-HCTZ Combination Tablet | Losartan Tablet + HCTZ Capsule
Number analyzed (Participants) | 20 | 20
ng*hr/mL | 462.08 (144.72) | 499.90 (133.46)
Statistical Analysis 1: Comparison: Losartan-HCTZ Combination Tablet vs Losartan Tablet + HCTZ Capsule; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence Bounds of (0.80, 1.25); Least-Squares Mean Ratio = 0.924, 90% CI [0.825 to 1.035]

4. Primary Outcome: Peak Plasma Concentration (Cmax) of HCTZ Following Single Dose Administration of Losartan/HCTZ or Losartan and HCTZ
Description: Peak Plasma Concentration (Cmax), or maximal concentration of drug following dosing
Time Frame: 30 Hours Post Dose
Population: Pharmacokinetic (PK) results were based on data from the 20 subjects who had blood drawn for the HCTZ assay. These 20 subjects were selected as the first 10 subjects from each treatment sequence who completed both periods of the study.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Losartan-HCTZ Combination Tablet | Losartan Tablet + HCTZ Capsule
Number analyzed (Participants) | 20 | 20
ng/mL | 76.15 (39.55) | 81.76 (31.05)
Statistical Analysis 1: Comparison: Losartan-HCTZ Combination Tablet vs Losartan Tablet + HCTZ Capsule; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Equivalence Bounds of (0.80, 1.25); Least-Squares Mean Ratio = 0.931, 90% CI [0.836 to 1.037]

ADVERSE EVENTS:
Description: Serious Adverse Events are reported by treatment group (Combination/Tablet+Capsule [N=38] or Tablet+Capsule/Combination [N=39]). For Other Adverse Events, the Combination/Tablet+Capsule group includes all subjects who received Combination Tablet (N=76) and the Tablet+Capsule/Combination group includes all subjects who received Tablet+Capsule (N=77)
Groups:
- Losartan Tablet +HCTZ Capsule/Losartan-HCTZ Combination Tablet: losartan 100 mg tablet + hydrochlorothiazide (HCTZ) 12.5 mg capsule then a single dose losartan 100 mg and HCTZ 12.5 mg combination tablet
Arm/Group | Losartan-HCTZ Combination Tablet/Losartan Tablet +HCTZ Capsule | Losartan Tablet +HCTZ Capsule/Losartan-HCTZ Combination Tablet
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 12/76 | 10/77
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losartan-HCTZ Combination Tablet/Losartan Tablet +HCTZ Capsule (N=76) | Losartan Tablet +HCTZ Capsule/Losartan-HCTZ Combination Tablet (N=77)
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 3
Headache (Nervous system disorders) | 8 | 6

LIMITATIONS AND CAVEATS:
PK analyses included complete data from 75 subjects. 3 losartan/E-3174 concentrations from 3 different subjects were excluded from analyses due to gross deviations; 75 minutes-Treatment B, 75 minutes-Treatment A, & 15 minutes-Treatment A.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.